CLINICAL TRIAL: NCT07083024
Title: Infection, Prevention and Control: A Multifaceted Approach to Preventing Hospital Acquired Infections Principal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Monakshi Sawhney, Associate Professor, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6040709
Record Dates: First submitted 2025-05-26; First posted 2025-07-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Infection Prevention
Keywords: education; nursing students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual education (Other): This is the baseline knowledge participants have
  Interventions: Behavioral: infection control education

INTERVENTIONS:
Behavioral: infection control education — This intervention includes a lecture, hands on practice and identifying IPAC practices in videos

SUMMARY:
Decreasing infections that occur when a person is hospitalized requires effective infection prevention and control (IPAC) practices. Lectures regarding IPAC as a way to provide education may not be effective for nursing students' learning. Other ways of educating nursing students is need. Therefore, the The aim of this study is to evaluate an alternative format of education that includes lectures, hands-on practice, and video scenarios.

Methods: This study uses a quasi-experimental design. Nursing students completing their final year of a Baccalaureate of Nursing program were included. The students attended a IPAC education session that included a lecture, hands-on practice, and a review of video scenarios. After the education session, knowledge was assessed using the post-test and videos related questions answered to demonstrate their ability to identify IPAC practices and lapses.

DETAILED DESCRIPTION:
In Canada, Health care associated infections affect more than 200,000 patients each year in Canada. The primary route of transmission of nosocomial pathogens are healthcare workers' hands and a secondary contributor to the transmission of pathogens within the hospital setting is the environment itself. The transmission of pathogens from health care workers and the environment to patients can be reduced through the use of routine infection prevention and control (IPAC) practices including completing a risk assessment, hand hygiene, controlling the environment (disinfecting equipment and surfaces), and the proper use of Personal Protective Equipment (PPE). All healthcare workers are responsible for implementing practices to reduce the spread of infection, including nursing students.

Nurses and nursing students are frequently exposed to blood and bodily fluids, emphasizing the importance of proper IPAC practices. Knowledge regarding IPAC practices varies from satisfactory to disappointing and even when nursing students have the correct knowledge they report rarely performing hand hygiene prior to non-invasive procedures There is a need to develop and implement multi-modal teaching strategies that improve the students' theoretical knowledge of IPAC and allow them to apply these concepts in an educational setting prior to implementing them within the clinical environment.

Different educational modalities including self-guided resources, synchronous teaching, or online modules can be used to provide theoretical nursing knowledge. However, to actively engage students with knowledge through practical application and hands-on experiences. To help bridge the gap between theoretical knowledge and application prior to clinical exposure, various teaching modalities have been proposed. This includes structured education programs, virtual simulation, interactive computer modules and simulated practice. Studies that have implemented these innovative teaching methodologies have demonstrated encouraging results related to IPAC practices.

An improvement in knowledge has been demonstrated in studies with nursing students after the addition of interactive and experiential learning to their didactic lessons. They also reported greater satisfaction with lessons when hands-on modalities allow for decision making without the risk of harm, allow engagement with a hospital-like environment, and reviews materials repeatedly In addition, despite having appropriate education, leadership and environmental cues heavily influence a student's implementation of IPAC practices. Students were more likely to forego the use of PPE when they noticed nurses in the clinical environment were not engaging in standard precautions. Therefore, it is essential to rethink how IPAC practices can be fully integrated into nursing student's routine practices to help mitigate the influence of what they witness in the clinical setting. Although there is a benefit to mixed modality teaching strategies, there is a gap in the literature regarding the effectiveness of an in-class mixed-modality educational session that combines didactic, hands-on practice, and videos on IPAC knowledge.

Aim The aim of this study is to evaluate the effectiveness the effectiveness of an innovative educational session that included didactic education intermingled with hands-on practice, and video scenarios on or final year nursing students' knowledge regarding the key steps in the prevention and control of the spread of infections. This study examined the following questions: for final year nursing students, what is the effect of an innovative IPAC education intervention on (a) change in knowledge regarding IPAC practices and (b) the ability to correctly identify errors in IPAC practices.

Methods This quasi experimental study utilizes a pre-test post-test design with nursing students enrolled in their final practicum at a University in Southern Ontario, Canada. Queen's University Research Ethics Board approval (HSREB# 6038157) was obtained prior to implementing this study.

Sample Final year Baccalaureate of Nursing Science (BNSc) students who were completing their final clinical placement students were invited to participate 24 hours prior to the education session during their regularly scheduled class time. Recruitment was completed by a member of the research team (a Master of Nursing Science student) and did not teach these students or determine their grades. All students were informed that participation in this study was voluntary and anonymous. The course instructor and the members of the research team would not be able to identify if they decided to participate in this study. Students were informed that if they decided not to participate in the study there would be no impact to grades or student success. Students who agreed to participate in this study completed an online consent form and completed a demographic questionnaire, and a pre-test to examine their baseline IPAC knowledge.

Setting The intervention took place during regular class time. All final year BScN students enrolled in the integrated practicum course participated in the IPAC education session, even if they did not participate in the study component.

Intervention

The intervention included an innovative IPAC education session that included didactic education intermingled with hands-on practice, and video scenarios. The IPAC education session was delivered over 2.5 hours and featured didactic education, hands-on practice, and videos scenarios of nurses in a simulated practice setting. The education session was grounded in information available from Public Health Ontario, Health Canada, and the World Health Organization. The video scenarios were developed by the research team and featured common nursing practices delivered in a hospital setting. During the education session the following concepts were explored:

1. the 'Chain of Infection' which highlights how infectious agents (viruses, bacteria, and fungi) are transmitted from person to person;
2. how to break the "Chain of Infection;"
3. effective hand hygiene;
4. the use of personal protective equipment (PPE), including masks;
5. cleaning versus disinfecting, and wet contact time of disinfectant agents. After each concept was introduced, all students completed a hands-on activity including a group hand hygiene exercise, donning and doffing gown, gloves and mask, and using two different disinfectant wipes (Lysol© = 4 minute wet contact time, and Oxivir TB© = 1 minute wet contact time) to disinfect a table and adhere to the wet contact time. Following the education session, video scenarios were used to engage the students in practice of identifying correct and incorrect IPAC practices. Students watched four videos, see Table 3 for a description of the video scenes.

Following the education session, the students who consented to participate in this study completed questions asking them to identify the correct and incorrect IPAC practices in each of the videos, and complete a post-test to evaluate the students' post-education session knowledge and potential practice change.

Outcome Measures Demographic information, including if students have completed past infection control education (in person or virtual), and if they have cared for patients who are under isolation precautions will be collected. Students will also complete the WHO Hand Hygiene Knowledge Questionnaire for Health-Care Workers. It includes 26 questions, and it is scored by summing the total number of correct answers. It has been used with practicing nurses working in a hospital setting and with nursing and medical students. The questionnaire has demonstrated a high reliability (α = 0.843).

Participants were also asked to report on their hand hygiene intentions and cleaning and disinfecting intention. These were measured using the Declarative Intention of Hand Hygiene Behavior and the Knowledge and Attitudes Regarding Hand Hygiene and Environmental Cleaning/Disinfecting. The Declarative Intention of Hand Hygiene Behavior and the Knowledge and Attitudes Regarding Hand Hygiene is based on the WHO four moments of hand hygiene. It includes 13 items which are recorded on a Likert scale that includes the options of 'never or very rarely'; 'sometimes'; or 'quite often or always.' The Knowledge and Attitudes Regarding Hand Hygiene and Environmental Cleaning/Disinfecting includes 10 items which are recorded on a Likert scale that includes the options of 'completely disagree'; 'somewhat agree'; and 'completely agree" Data Collection All data, including the consent forms were anonymous and were collected using a web-based survey tool (Qualtrics©). The anonymous web-based links to the consent and pre-test and post-test questionnaires were posted on the final year nursing students' course page. All students had access to these links, and had the choice to participate in this study. The course professor had no knowledge regarding which students agreed to participate.

Data Analysis Data was analyzed using Statistical Package for the Social Sciences (SPSS© version 29). Demographic information was analyzed using means, standard deviations, and frequencies. The frequencies were calculated for the Declarative intention of hand hygiene behavior and the Knowledge and Attitudes Regarding Hand Hygiene and Environmental Cleaning/Disinfecting questions. A Kolmogorov-Smirnov test indicated that the results from the pre-test (df = 56, p = 0.16) and the post-test (df = 56, p < 0.01) for the WHO Hand Hygiene Questionnaire (World Health Organization, 2009) did not follow a normal distribution therefore the median pre-test and post-test scores were calculated. To examine if there were any significant changes in knowledge from the pre-test and post-test results a Wilcoxon Signed Rank Test was used.

ELIGIBILITY:
Inclusion Criteria:

- Final year Baccalaureate of Nursing Science (BNSc) students

Exclusion Criteria:

- Students not enrolled in the BNSc program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
WHO Hand Hygiene Knowledge Questionnaire for Health-Care Workers (World Health Organization, 2009) | Day 1
  It includes 26 questions, and it is scored by summing the total number of correct answers. It has been used with practicing nurses working in a hospital setting and with nursing and medical students. The questionnaire has demonstrated a high reliability (α = 0.843).

SECONDARY OUTCOMES:
Declarative Intention of Hand Hygiene Behavior and the Knowledge and Attitudes Regarding Hand Hygiene and Environmental Cleaning/Disinfecting | Day 1
  The Declarative Intention of Hand Hygiene Behavior and the Knowledge and Attitudes Regarding Hand Hygiene is based on the WHO four moments of hand hygiene. It includes 13 items which are recorded on a Likert scale that includes the options of 'never or very rarely'; 'sometimes'; or 'quite often or always.' The Knowledge and Attitudes Regarding Hand Hygiene and Environmental Cleaning/Disinfecting includes 10 items which are recorded on a Likert scale that includes the options of 'completely disagree'; 'somewhat agree'; and 'completely agree"

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada